CLINICAL TRIAL: NCT03488589
Title: Hepatitis E Virus Infection Among Patients With Acute Non-A, Non-B, Non-C Hepatitis in Al-Rajhy University Hospital for Liver
Brief Title: HEV in Patients With Acute Non-A, Non-B, Non-C Hepatitis in Al-Rajhy University Hospital for Liver
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Abdel Rahman (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Abdel Rahman, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Assiut2018
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis E
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum samples for HEV RNA PCR — serum samples HEV RNA PCR

SUMMARY:
Hepatitis E is the fifth known human viral hepatitis and is probably the most common cause of acute viral hepatitis in the world. The incidence of acute hepatitis E is estimated at 3 million human cases per year worldwide, with around 70,000 deaths. Most cases occur in endemic countries, but the number of cases in low-endemic areas has increased. HEV seroprevalence is high in developing countries, such as India and Southeast Asia, ranging from 27-80%. Acute disease mortality is 1-4%, with risk being higher in pregnant women and immunodeficient patients.

The four more prevalent genotypes are allocated into two groups. Epidemic hepatitis E includes genotypes 1 and 2, which are considered human viruses and have caused the epidemics of hepatitis. These forms are transmitted mainly by contaminated water and the fecal-oral route. endemic hepatitis E includes genotypes 3 and 4, which are considered swine viruses (common in domestic and wild pigs), capable of infecting humans as an accidental host and therefore considered zoonotics.

The course and clinical presentation of hepatitis E is highly variable. The detailed mechanisms that lead to the different clinical outcomes in hepatitis E are only partially understood. It is known that both viral factors (genotype and dose of inoculum) and host factors (presence of previous liver disease, pregnancy and distinct genetic polymorphisms) determine the course of infection. In most cases, hepatitis E causes self-limited illness, lasting from a few days to weeks, with an average of 4-6 weeks. However, in developed countries it can cause chronic disease with rapid progression to cirrhosis, especially in patients who are transplanted, have hematological malignancies requiring chemotherapy, or have infection with HIV.

Hepatitis E is an underdiagnosed disease, partly due to the use of serological tests with low sensitivity. Diagnosis can be made indirectly by detecting antibodies against HEV in the serum, or directly by detecting the genome of the virus in blood or other body fluids. The tests for anti-hepatitis E antibody screening are commercially available, but none of them has been approved by the Food and Drug Administration (FDA). Unfortunately, the sensitivity and specificity of these tests vary greatly and this could explain the discrepancies in rates of anti-hepatitis E antibodies published for the various populations studied. The tests for viral RNA in serum and feces are confirmatory, but still experimental.

ELIGIBILITY:
Inclusion Criteria:

* • Patients have clinical diagnosis of acute viral hepatitis as (recent onset of nausea, fever, fatigue, abdominal pain , hepatomegaly and abnormal transaminases (at least 2 fold higher than the upper normal level))

  * Post-transplant acute hepatitis

Exclusion Criteria:

* hepatitis A, B and C patients
* autoimmune hepatitis
* Alcoholism
* Treatment with hepatotoxic drugs
* Biliary disease
* Infection with CMV or EBV
* Taken ribavirin therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients fulfilling the inclusion criteria of acute hepatitis either admitted to Al-Rajhi University hospital for liver,visiting Al-Rajhy university hospital outpatient clinics for gastroentrology and hepatology or consultations from other departments at Assiut University hospitals
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
HEV incidence estimation among acute hepatitis patients | 1-2 years
  in our university hospital HEV is underestimated due to the lack of laboratory investigation of it . so, by this study we aim to estimate the number of affected cases with HEV infection among symptomatic patients with acute hepatitis.

SECONDARY OUTCOMES:
Detection of Hepatitis E viral nucleic acid in stool and serum | 1-2 years
  Detection of Hepatitis E viral nucleic acid in stool and serum of acute non- A, B or C hepatitis patients and compare between the viral load in both samples. and according the results we can recommend the preferred sample type to be used later for detection of the virus .

OTHER OUTCOMES:
medical recommendation | 1-2 years
  if our study found high incidence of HEV among patients with acute hepatitis , we can then recommend (with evidence) adding Acute HEV infection testing modalities as a routine investigation to AL-Rajhy hospital protocols in managing Acute hepatitis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Reda, professor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code